CLINICAL TRIAL: NCT06903728
Title: National forsøgsordning Med Glukosesensorer Til Type 2-diabetes: Glukosesensorer Til Gravide Med Type 2-diabetes
Brief Title: National Trial of CGM in Pregnant Women With Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Steno Diabetes Center Odense (Other); Steno Diabetes Center Copenhagen (Other); Steno Diabetes Center Aarhus (SDCA), Aarhus University Hospital (Unknown); Steno Diabetes Center Nordjylland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGM til gravide med T2D
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes; Pregnancy
Keywords: CGM in type 2 diabetes; CGM in pregnancy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Sensor use (Experimental): Participants are given a sensor to use during pregnancy until 4-6 weeks post partum
  Interventions: Device: continous glucose monitoring

INTERVENTIONS:
Device: continous glucose monitoring — Pregnant women with type 2 diabetes are given a sensor < week 14 of their pregnancy and will use it until 4-6 post partum. They will receive training in how to use the sensor, and support when needed.

SUMMARY:
The goal of this clinical trial is to evaluate the use of glucose sensors in pregnant women with type 2 diabetes to improve insulin regulation, pregnancy and birth outcomes, and enhance quality of life and satisfaction with treatment.

The main questions it aims to answer are:

* Does the use of glucose sensors during pregnancy lead to a clinically significant reduction in HbA1c by 0.3% at 36 weeks gestation compared to the control group?
* Does the use of glucose sensors during pregnancy result in a clinically significant reduction in mean SD-score for birth weight deviation in newborns compared to the control group?

Researchers will compare the group of women using glucose sensors during pregnancy to a historical control group receiving routine care to see if the sensor improves pregnancy outcomes, glucose control, and birth weights.

Participants will:

* Use a glucose sensor from before 14 weeks of pregnancy until 4-6 weeks postpartum.
* Receive training on how to use the sensor and access ongoing support as needed.
* Have a follow-up appointment 4-6 weeks postpartum, including a consultation for advice on medical treatment and further management of diabetes after birth.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with type 2 diabetes
* attending one of the four centers for pregnancy and diabetes in Denmark
* 18 years old or above

Exclusion Criteria:

* gestationel age 14+0 or above
* ekspected birth after end of trial
* already using a continous glucose monitor (sensor)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c at end of pregnancy (week 36 of pregnancy) | baseline < week 14 of pregnancy, follow up week 36 of pregnancy
child birth weight SD-score | at time of birth

SECONDARY OUTCOMES:
TIR, TAR, TBR | from enrollment to 4-6 weeks post partum
  Percentage of time in time in range, time above range and time below range during their pregnancy.
Mean glucose | from enrollment to 4-6 weeks post partum
  Sensor specific data
Womens gestational wheight gain | from enrollment to birth
  weight gain during throughout pregnancy
Hypoglykemia among newborn | at time of birth
  Hypoglykemia among newborn
Pregnancy related complications | from enrollment to birth
  increased blood pressure and preeclampsia
Birth related complications | at time of birth
  c-section, early birth
Problem Areas in Diabetes (PAID) | Baseline, week 28, 4-6 weeks post partum
  Diabetes stress
World Health Organisation - Five Well-Being Index (WHO-5) | Baseline, week 28, 4-6 weeks post partum
  quality of life
12-Item Short-Form (SF12) | Baseline, week 28, 4-6 weeks post partum
  Health status
Patient Assessment of Cronic Illness Care (PACIC) | Baseline, week 28, 4-6 weeks post partum
  Satisfaction with care
Glucose Monitoring Satisfaction Survey (GMSS) | Baseline, week 28, 4-6 weeks post partum
  Satisfaction with method used for glucose measuring
Pregnancy Physical Activity Questionnaire (PPAQ-DK | Baseline, week 28
  Physical activity in pregnancy
Diet items from the National Danish Birth Cohort | Baseline, week 28
  Pregnancy specific questions related to diet

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: December 2025 and december 2026